CLINICAL TRIAL: NCT05317234
Title: Genetic Predisposition in Cerebral Palsy
Acronym: PREGENE PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL21_0849
Record Dates: First submitted 2022-03-22; First posted 2022-04-07 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Genetic predisposition; Neurodevelopmental disorder
MeSH Terms: conditions — Cerebral Palsy; Genetic Predisposition to Disease; Neurodevelopmental Disorders | interventions — Exome

STUDY DESIGN:
Intervention Model Description: Patients between 2 and 17 years old, born from 34 weeks' gestation, with a diagnosis of cerebral palsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- children with cerebral palsy (Experimental): Patients between 2 and 15 years old, born after 34 weeks' gestation, with a diagnosis of cerebral palsy.
  Interventions: Genetic: Whole-exome sequencing

INTERVENTIONS:
Genetic: Whole-exome sequencing — The whole-exome sequencing will be performed via a blood sample from a patient with a diagnosis of cerebral palsy.

SUMMARY:
Cerebral palsy (CP) is a major neurodevelopmental disorder with an estimated prevalence of approximately one in 500 children. It is characterised by permanent developmental disorders of movement and posture, responsible for activity limitations, caused by non-progressive damage to the brain of the fetus, newborn or infant during development. The neurobiological mechanisms involved in CP remain poorly understood, although the interruption of cerebral oxygen supply during pregnancy or at the time of delivery is classically considered to be the main factor causing neurodevelopmental sequelae. CP also occurs in full-term infants without a clearly identifiable etiology.

Data from the literature suggest the existence of other pathophysiological processes than only acquired brain lesions related to pregnancy and delivery, such as genetic or epigenetic factors. According to some research teams, nearly one third of CP could have a genetic cause or could be favoured by genetic variants.

Preliminary research has made significant progress in revealing unusual copy number variants and/or mutations in single genes in children with CP. Several of the identified genes are involved in neurodevelopment and neuronal connectivity. Nevertheless, the identification of these abnormalities in CP may contribute to a better understanding of the pathophysiology of this complex and multifactorial disorder. It could also shed new light on the analysis of medico-legal files and bring encouraging perspectives by targeting new therapeutic interventions.

The main hypothesis is that a certain number of cerebral palsies are related to - or favoured by - genetic abnormalities that we will search for with genetic screening tests.

ELIGIBILITY:
Inclusion Criteria:

* Child between 2 and 15 years old with a clinical diagnostic of cerebral paralysis with unilateral or bilateral somatic involvement
* Child born from 34 SA
* Agreement of the legal representatives for the genetic study
* Both parents available for a parental genetic study (if detection of class 3 variant)
* Affiliation to the social security system

Exclusion Criteria:

* Genetic syndrome identified or malformative or infectious etiologies identified
* Neonatal encephalopathy criteria in a clear obstetrical etiological context responsible for major perinatal anoxia with Sarnat 2 or 3
* Unilateral motor disorders in perinatal stroke of identified etiology (coagulation anomaly)

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2028-03-08 (Estimated); Study Completion 2028-03-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom a significant genetic variant was identified on the exome by the High-throughput sequencing technique after comparison with the databases of human polymorphisms and pathogenic variants up to date during the analysis. | Until the end of study, an average of 4.5 years
  Are considered positive for a significant genetic variant, patients for whom a or several class 4 or 5 variants have been identified, and explain the phenotype of pc. Genetic variants will be classified according to the recommendations of the American College of Genetics Medical (ACMG: American College of Medical Genetics) from 1 to 5.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de Médecine Physique et Réadaptation Pédiatrique - Hôpital Femme-Mère-Enfant, Bron
  - Service de médecine physique et réadaptative pédiatrique, Pôle pédiatrie-Génétique - Hôpital Couple-Enfant, Grenoble